CLINICAL TRIAL: NCT01923285
Title: A Prospective, Randomized, Multi-Center, Controlled Clinical Trial to Assess the Safety and Efficacy of the Spinal Modulation™ AXIUM™ Neurostimulator System in the Treatment of Chronic Pain (ACCURATE Trial)
Brief Title: A Safety and Effectiveness Trial of Spinal Cord Stimulation of the Dorsal Root Ganglion for Chronic Lower Limb Pain
Acronym: ACCURATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-SMI-2012
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Chronic Lower Limb Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AXIUM Neurostimulator System (Experimental): The AXIUM Neurostimulator System is an investigational spinal cord stimulation device that is designed to stimulate the dorsal root ganglion (DRG) of the spine located on the back surface of the spinal cord where nerves exit the backbone. The device has 2 parts that are placed surgically (implanted) : 1) a pulse generator which is placed under the skin in the buttocks or abdomen, and 2) up to four wires (leads) that have one end attached to the pulse generator, and the other end secured to the tissue near the target treatment area.
  Interventions: Device: AXIUM Neurostimulator System
- Control Spinal Cord Stimulation Device (Active Comparator): The Control Spinal Cord Stimulation Device is a commercially available spinal cord stimulator indicated for the treatment of chronic lower limb pain.
  Interventions: Device: Control Spinal Cord Stimulation Device

INTERVENTIONS:
Device: AXIUM Neurostimulator System
  Other Names: DRG Stimulation
  Arms: AXIUM Neurostimulator System
Device: Control Spinal Cord Stimulation Device
  Other Names: SCS
  Arms: Control Spinal Cord Stimulation Device

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the AXIUM Neurostimulator System for the treatment of chronic lower limb pain in persons diagnosed with Complex Regional Pain Syndrome (CRPS) or Peripheral Causalgia (PC).

DETAILED DESCRIPTION:
The ACCURATE study is a prospective, randomized, controlled, multicenter clinical trial designed to assess the safety and efficacy of the Spinal Modulation Axium Neurostimulator System as an aid in the management of chronic, intractable pain of the lower limbs, including unilateral or bilateral pain associated with one of the following conditions: Complex Regional Pain Syndrome (CRPS) or Peripheral Causalgia (also referred to as CRPS Type II).

Enrolled subjects were diagnoses with CRPS or peripheral causalgia; experienced pain for at least six months; and failed to achieve adequate pain relief from at least two prior pharmacologic treatments.

All subjects had a temporary trial neurostimulator (TNS). If the subject was a treatment success at the end of TNS they were scheduled for the fully implantable neurostimulator (INS) implant procedure. If not, subjects were exited from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between the ages of 22 and 75 years
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Subject has chronic, intractable pain of the lower limb(s) for at least 6 months
4. Subjects are diagnosed with complex regional pain syndrome (CRPS) and/or peripheral causalgia
5. Subjects have a minimum Visual Analog Scale (VAS) greater than or equal to 60 mm in the area of greatest pain in the lower limbs.
6. Subject has failed to achieve adequate pain relief from at least 2 prior pharmacologic treatments from at least 2 different drugs classes
7. Subject has had stable neurologic function in the past 30 days
8. In the opinion of the Investigator, the subject is psychologically appropriate for the implantation of an active implantable medical device
9. Subject is able to provide written informed consent

Exclusion Criteria:

1. Back pain is the greatest region of pain as measured on the baseline VAS.
2. Female subject of childbearing potential is pregnant/nursing, plans to become pregnant or is unwilling to use approved birth control
3. Subject has exhibited escalating or changing pain condition within the past 30 days as evidenced by Investigator examination
4. Subject is currently involved in medically related litigation, including workers compensation
5. Subject has had corticosteroid therapy at an intended site of stimulation within the past 30 days
6. Subject's pain medication(s) dosage(s) are not stable for at least 30 days
7. Subject has had radiofrequency treatment of an intended target Dorsal Root Ganglion within the past 3 months
8. Subject has previously failed spinal cord stimulation therapy
9. Subject currently has an active implantable device including implantable cardioverter defibrillator, pacemaker, spinal cord stimulator or intrathecal drug pump or subject requires magnetic resonance imaging (MRIs) or diathermy
10. Subject has pain only within a cervical distribution
11. Subject has cognitive, physical or sensory impairment that, in the opinion of the Investigator, may limit their ability to operate the device
12. Subject currently has an indwelling device that may pose an increased risk of infection
13. Subject currently has an active systemic infection.
14. Subject has, in the opinion of the investigator, a medical comorbidity that contraindicates placement of an active medical device
15. Subject has participated in another clinical investigation within 30 days
16. Subject has a coagulation disorder or uses anticoagulants that, in the opinion of the Investigator, precludes participation
17. Subject has been diagnosed with cancer in the past 2 years
18. Imaging (MRI, CT, x-ray) findings within the last 12 months that, in the Investigator's opinion, contraindicates lead placement
19. Subject is a prisoner

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Capobianco, PhD, Study Director — Abbott
Locations (22):
- United States (22):
  - HOPE Research - TPC, Phoenix, Arizona
  - Pain Clinic of Monterey Bay, Aptos, California
  - Coastal Pain Research, Carlsbad, California
  - Neurovations, Inc., Napa, California
  - Newport Beach Headache and Pain, Newport Beach, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Orthopaedic Pain Specialists, Santa Monica, California
  - IPM Medical Group, Inc., Walnut Creek, California
  - Florida Pain Institute, Merritt Island, Florida
  - Holy Cross Hospital Orthopedic Institute, Oakland Park, Florida
  - Drug Studies of America, Marietta, Georgia
  - Comprehensive Pain and Rehabilitation, Pascagoula, Mississippi
  - Pain Management Associates, Independence, Missouri
  - HOPE Research - LVSP, Las Vegas, Nevada
  - Premier Pain Center, Shrewsbury, New Jersey
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Southeastern Spine Institute, Mt. Pleasant, South Carolina
  - Houston Pain Centers, Houston, Texas
  - Center for Pain Relief, Charleston, West Virginia
  - Center for Pain Relief Tri-State, Huntington, West Virginia

REFERENCES:
- [Derived] Levy RM, Mekhail N, Kramer J, Poree L, Amirdelfan K, Grigsby E, Staats P, Burton AW, Burgher AH, Scowcroft J, Golovac S, Kapural L, Paicius R, Pope J, Samuel S, McRoberts WP, Schaufele M, Kent AR, Raza A, Deer TR. Therapy Habituation at 12 Months: Spinal Cord Stimulation Versus Dorsal Root Ganglion Stimulation for Complex Regional Pain Syndrome Type I and II. J Pain. 2020 Mar-Apr;21(3-4):399-408. doi: 10.1016/j.jpain.2019.08.005. Epub 2019 Sep 5. PMID 31494275

RESULTS

PARTICIPANT FLOW:
Groups:
- AXIUM Neurostimulator System: The AXIUM Neurostimulator System is an investigational spinal cord stimulation device that is designed to stimulate the dorsal root ganglion (DRG) of the spine located on the back surface of the spinal cord where nerves exit the backbone. The device has 2 parts that are placed surgically (implanted) : 1) a pulse generator which is placed under the skin in the buttocks or abdomen, and 2) up to four wires (leads) that have one end attached to the pulse generator, and the other end secured to the tissue near the target treatment area.
  AXIUM Neurostimulator System
- Control Spinal Cord Stimulation Device: The Control Spinal Cord Stimulation Device is a commercially available spinal cord stimulator indicated for the treatment of chronic lower limb pain.
  Control Spinal Cord Stimulation Device
Period: Overall Study
Arm/Group | AXIUM Neurostimulator System | Control Spinal Cord Stimulation Device
Started | 76 | 76
Modified Intent-to-treat (6 subjects excluded from MITT (withdrew prior to trial phase): Axium N = 3, Control N = 3) | 73 | 73
Completed | 69 | 70
Not Completed | 7 | 6
Not completed — Withdrawal by Subject | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AXIUM Neurostimulator System | Control Spinal Cord Stimulation Device | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Median (Full Range); unit: Years] | 53.2 [23.9 to 75.8] | 53 [25.4 to 75.9] | 53 [23.9 to 75.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 37 | 39 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Black or African American | 2 | 3 | 5
  Race: Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Race: White | 72 | 70 | 142
  Race: Other | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 8 | 12
  Ethnicity: Not Hispanic or Latino | 72 | 68 | 140
Region of Enrollment [Number; unit: participants]
  United States | 76 | 76 | 152
Body Mass Index (BMI) [Median (Full Range); unit: kg/m2] | 29.9 [16.9 to 54.0] | 27.9 [17.4 to 44.6] | 29.9 [16.9 to 54.0]
Primary Diagnosis [Count of Participants; unit: Participants]
  Complex Regional Pain Syndrome | 44 | 43 | 87
  Peripheral Causalgia | 32 | 33 | 65
Duration of Lower Limb Pain [Median (Full Range); unit: Years] | 5.0 [1.0 to 39.0] | 4.5 [0.7 to 51.0] | 5.0 [0.7 to 51.0]
Primary Region of Pain [Count of Participants; unit: Participants]
  Region 2 - Right Groin | 4 | 2 | 6
  Region 3 - Left Groin | 4 | 7 | 11
  Region 4 - Right Buttock | 2 | 2 | 4
  Region 5 - Left Buttock | 1 | 2 | 3
  Region 6 - Right Leg | 14 | 16 | 30
  Region 7 - Left Leg | 8 | 11 | 19
  Region 8 - Right Foot | 21 | 19 | 40
  Region 9 - Left Foot | 22 | 17 | 39

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Endpoint - Treatment Success
Description: Treatment Success is defined as at least 50% lower limb pain relief (VAS score reduction) at the end of trial phase, received at least 50% lower limb pain relief at the 3-month visit post implant, and the absence of a stimulation related neurological deficit. Pain scores were measured using Visual Analog Scale (VAS). The VAS score ranges from 0-100 mm with a higher score indicating higher pain intensity ( 0 representing "No Pain" and 100 mm representing "Worst Imaginable Pain").
Time Frame: 3 months
Population: Subjects excluded since they do not have evaluable data: Axium=4, Control=3. Seven subjects in the MITT analysis have no evaluable data for the study endpoints due to withdrawing prior to the 3-mo study visit and did not meeting criteria for treatment failure/success upon study exit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AXIUM Neurostimulator System | Control Spinal Cord Stimulation Device
Number analyzed (Participants) | 69 | 70
percentage of subjects | 81.2 [69.9 to 89.6] | 55.7 [43.3 to 67.6]
Statistical Analysis 1: Comparison: AXIUM Neurostimulator System vs Control Spinal Cord Stimulation Device; The primary hypothesis tested was: H0: p1 ≤ p0 - δ vs. H1: p1> p0 - δ, where p0 is the success rate in the Control group, p1 is the success rate in the Axium group, and δ is the non-inferiority margin, which is pre-specified at 10%. If non-inferiority is achieved at a one-sided alpha of 0.05, a one-sided superiority test is performed at the significance level of 0.025; Test type: Non-Inferiority — The non-inferiority margin, which is pre-specified at 10%. If non-inferiority is achieved at a one-sided alpha of 0.05, a one-sided superiority test is performed at the significance level of 0.025; p < 0.0001, Chi-squared — The non-inferiority margin, which is pre-specified at 10%. If non-inferiority is achieved at a one-sided alpha of 0.05, a one-sided superiority test is performed at the significance level of 0.025
Statistical Analysis 2: Comparison: AXIUM Neurostimulator System vs Control Spinal Cord Stimulation Device; The primary hypothesis tested was: H0: p1 ≤ p0 - δ vs. H1: p1> p0 - δ, where p0 is the success rate in the Control group, p1 is the success rate in the Axium group, and δ is the non-inferiority margin, which is pre-specified at 10%; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0004, Chi-squared

2. Secondary Outcome: Positional Effects on Paresthesia Intensities
Description: Positional effects on paresthesia intensities at 3 months in the Control group versus the Treatment Group. This endpoint will compare the difference in paresthesia scores upright and supine between the AXIUM and Control groups. Paresthesia intensity was rated by subjects using a paresthesia intensity rating scale. Subjects rated the intensity of their perception of paresthesia, while upright and supine, on an 11-point numeric rating scale from 0 representing "No feeling" to 10 "Very intense." Perceived paresthesia intensity difference between supine and upright positions was calculated and averaged across each group.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AXIUM Neurostimulator System | Control Spinal Cord Stimulation Device
Number analyzed (Participants) | 56 | 53
score on a scale | -0.1 (1.6) | 1.8 (3.0)
Statistical Analysis 1: Comparison: AXIUM Neurostimulator System vs Control Spinal Cord Stimulation Device; Secondary endpoint compared the mean differences in upright and supine paresthesia scores between the Axium and Control groups at three months post INS implant. This endpoint was evaluated at a two-sided significance level of 0.05. The primary hypothesis tested was: H0: μ0- μ1≤0 vs. H1: μ0- μ1>0 where μ0 is the mean difference in paresthesia intensities in the Control group and μ1 is the mean difference in the Axium group; Test type: Other — Comparison of the mean difference. Difference in intensities is calculated as the supine paresthesia intensity minus the upright paresthesia intensity; p < 0.0001, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 1.9, 95% CI 2-sided [1.0 to 2.8] — Difference in paresthesia intensities is calculated as the supine paresthesia score minus the upright paresthesia score for each subject

3. Other Pre Specified Outcome: Primary Composite Endpoint - Treatment Success for Only Those Subjects With a Permanent Implant
Description: Treatment Success is defined as a reduction in pain score greater than or equal to 50 percent and the absence of a stimulation related neurological deficit. Pain scores were measured using Visual Analog Scale (VAS). The VAS score ranges from 0-100 mm with a higher score indicating higher pain intensity ( 0 representing "No Pain" and 100 mm representing "Worst Imaginable Pain").
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AXIUM Neurostimulator System | Control Spinal Cord Stimulation Device
Number analyzed (Participants) | 61 | 54
percentage of subjects | 93.3 [83.3 to 98.2] | 72.2 [58.4 to 83.5]
Statistical Analysis 1: Comparison: AXIUM Neurostimulator System vs Control Spinal Cord Stimulation Device; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — If non-inferiority is achieved at a one-sided alpha of 0.05, a one-sided superiority test is performed at the significance level of 0.025; p < 0.0001, Chi-squared
Statistical Analysis 2: Comparison: AXIUM Neurostimulator System vs Control Spinal Cord Stimulation Device; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.0047, Chi-squared

4. Other Pre Specified Outcome: Primary Composite Endpoint - Treatment Success for Only Those Subjects With a Permanent Implant
Description: as for outcome 3
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AXIUM Neurostimulator System | Control Spinal Cord Stimulation Device
Number analyzed (Participants) | 57 | 51
percentage of subjects | 86 [74.2 to 93.7] | 68.6 [54.1 to 80.9]
Statistical Analysis 1: Comparison: AXIUM Neurostimulator System vs Control Spinal Cord Stimulation Device; [analysis description as in outcome 1, analysis 2]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; p = 0.0003, Non-inferiority

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of subject enrollment through completion of study follow-up or early discontinuation, whichever occured first, an average of 1 year.
Description: An AE is an untoward medical occurrence in a patient or subject implanted with a study device whether or not the event has causal relationship to the device; can be any unfavorable or unintended sign, symptom, disease temporally associated with device use. An AE is serious if it meets any of the following: immediately life threatening, results in disability, requires invasive intervention to preclude permanent impairment or death, results in or prolongs hospitalization, or results in death.
Arm/Group | AXIUM Neurostimulator System | Control Spinal Cord Stimulation Device
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 8/76 | 15/76
Other Adverse Events (participants affected / at risk) | 5/76 | 5/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIUM Neurostimulator System (N=76) | Control Spinal Cord Stimulation Device (N=76)
Abnormal blood chemistry (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lower extremity/bilateral leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Substance relayed disorder/overdose or withdrawal (Psychiatric disorders) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Injury/ADL (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Joint or muscle surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac valve (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Dermatologic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eyes or ears or nose or throat (General disorders) | 0 (0) | 1 (1)
Cholecystectomy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Systemic infection or general (Infections and infestations) | 0 (0) | 1 (1)
Fall injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Trunk or rib pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXIUM Neurostimulator System (N=76) | Control Spinal Cord Stimulation Device (N=76)
Side effect/Procedure medication (General disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No